CLINICAL TRIAL: NCT04010656
Title: Optimization of Spontaneous Trial of Void: a Prospective Cohort Study
Brief Title: Optimization of Spontaneous Postoperative Trial of Void Among Women
Acronym: OPTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: American Urogynecologic Society (Other); American Association of Gynecologic Laparoscopists (Other)
Responsible Party: Principal Investigator, Anne Cooper, MD, Assistant Professor of Urogynecology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WIH IRB 1145237
Record Dates: First submitted 2019-02-19; First posted 2019-07-08 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Urinary Retention Postoperative; Voiding Disorders
Keywords: Urogynecologic surgery; Urinary retention postoperative

STUDY DESIGN:
Intervention Model Description: Subjects will be taught to perform self-catheterization prior to prolapse repair or incontinence surgery; voiding data will be collected on the participant's first void after surgery. Participants will be discharged home to perform self-catheterization until post-void residual is less than half the volume voided on 2 sequential voids to assess actual voiding function, and this data will be used to calculate the diagnostic accuracy of pre-determined combinations of the TOV parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PVR-based home self-catheterization (Experimental): Patients will learn to self-catheterize preoperatively prior to urogynecology surgery requiring trial of void. First post-operative void will be used to collect basic information about voiding function. All participants will leave the hospital and self-catheterize until they achieve two sequential voids with post-void residual (PVR) less than half the volume voided. The cases of urinary retention captured with abnormal PVR will be used to compare the diagnostic accuracy of several commonly-used, pre-defined parameters for trial of void.
  Interventions: Procedure: PVR-based self-catheterization

INTERVENTIONS:
Procedure: PVR-based self-catheterization — Home self-catheterization based on standard of care

SUMMARY:
Trial of void (TOV) is a diagnostic test performed on all women who undergo prolapse repair or incontinence surgery, due to the importance of diagnosing postoperative urinary retention (POUR). Incidence of POUR may be as high as 62% in some studies. Timely and accurate diagnosis is important to avoid complications such as urinary tract infection, bladder overdistension, and permanent bladder injury. Despite the frequent use of TOV, there is no gold standard for the test, and it likely has poor specificity, leading to discharge of more patients with catheter than required. This prospective cohort study will seek to establish evidence-based optimal parameters for spontaneous trial of void, a TOV modality that has merit for further evaluation given lower theoretical risk of urinary tract infection.

DETAILED DESCRIPTION:
Patients will learn to perform self-catheterization ('clean intermittent catheterization', or CIC) preoperatively; after surgery, the investigators will collect a range of voiding parameters used during different TOV protocols (including minimum voided volume [MVV], post-void residual via bladder scanner [PVR], subjective force of urinary stream [sFOS]). Patients will discharge home to perform CIC until two sequential post-void residuals of less than half the volume voided have been achieved. The rate of voiding dysfunction and resulting PVRs will be used to compare the diagnostic accuracy of the perioperative voiding parameters to predict need to perform CIC and post-operative urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking women, age >18yo
* Scheduled for urogynecology procedure which will need post-operative trial of void (including pelvic organ prolapse and/or stress urinary incontinence repair), with plan for same-day discharge.

Exclusion Criteria:

* Unable or unwilling to perform self-catheterizatoin either by patient or willing family member
* Pre-existing voiding dysfunction defined as documented PVR > 200 mL
* Intraoperative urinary tract injury needing indwelling catheter on discharge
* Need for overnight admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative urinary retention | 24-72 hours postoperative
  Based on defined criteria
Diagnostic accuracy of trial of void parameters | First void postoperative (within 4 hours postop)
  Comparison of sensitivity, specificity, positive/negative predictive value of different trial of void parameters from first postoperative void, based on those used in the literature.

SECONDARY OUTCOMES:
Rate of post-operative and post-discharge urinary retention | 24-72 hours postoperative
  Based on post-void residual volume
Rate of post-operative urinary tract infection | 6 weeks postoperative
  UTI in first 6 weeks postoperative
Patient satisfaction with self-catheterization method via questionnaire | 2 weeks postoperative
  Novel questionnaire, 5 point Likert scale from "Very dissatisfied to Very satisfied"
Time to first void postoperative | 4 hours postoperative
  To assess time to spontaneous void after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Cooper, MD, MA, Principal Investigator — Dartmouth-Hitchcock Medical Center, Lebanon NH; Julia Shinnick, MD, Principal Investigator — Women & Infants Hospital, Providence RI
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorflinger A, Monga A. Voiding dysfunction. Curr Opin Obstet Gynecol. 2001 Oct;13(5):507-12. doi: 10.1097/00001703-200110000-00010. PMID 11547032
- [Background] Partoll LM. Efficacy of tension-free vaginal tape with other pelvic reconstructive surgery. Am J Obstet Gynecol. 2002 Jun;186(6):1292-5; discussion 1295-8. doi: 10.1067/mob.2002.123736. PMID 12066111
- [Background] Barber MD, Kleeman S, Karram MM, Paraiso MF, Walters MD, Vasavada S, Ellerkmann M. Transobturator tape compared with tension-free vaginal tape for the treatment of stress urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2008 Mar;111(3):611-21. doi: 10.1097/AOG.0b013e318162f22e. PMID 18310363
- [Background] Geller EJ. Prevention and management of postoperative urinary retention after urogynecologic surgery. Int J Womens Health. 2014 Aug 28;6:829-38. doi: 10.2147/IJWH.S55383. eCollection 2014. PMID 25210477
- [Background] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294
- [Background] de Souza GM, Costa WS, Bruschini H, Sampaio FJ. Morphological analysis of the acute effects of overdistension on the extracellular matrix of the rat urinary bladder wall. Ann Anat. 2004 Feb;186(1):55-9. doi: 10.1016/S0940-9602(04)80122-5. PMID 14994912
- [Background] Rosseland LA, Stubhaug A, Breivik H. Detecting postoperative urinary retention with an ultrasound scanner. Acta Anaesthesiol Scand. 2002 Mar;46(3):279-82. doi: 10.1034/j.1399-6576.2002.t01-1-460309.x. PMID 11939918
- [Background] Asimakopoulos AD, De Nunzio C, Kocjancic E, Tubaro A, Rosier PF, Finazzi-Agro E. Measurement of post-void residual urine. Neurourol Urodyn. 2016 Jan;35(1):55-7. doi: 10.1002/nau.22671. Epub 2014 Sep 22. PMID 25251215
- [Background] Wheeler TL 2nd, Richter HE, Greer WJ, Bowling CB, Redden DT, Varner RE. Predictors of success with postoperative voiding trials after a mid urethral sling procedure. J Urol. 2008 Feb;179(2):600-4. doi: 10.1016/j.juro.2007.09.080. Epub 2007 Dec 21. PMID 18082219
- [Background] Hakvoort RA, Dijkgraaf MG, Burger MP, Emanuel MH, Roovers JP. Predicting short-term urinary retention after vaginal prolapse surgery. Neurourol Urodyn. 2009;28(3):225-8. doi: 10.1002/nau.20636. PMID 19130599
- [Background] Ripperda CM, Kowalski JT, Chaudhry ZQ, Mahal AS, Lanzer J, Noor N, Good MM, Hynan LS, Jeppson PC, Rahn DD. Predictors of early postoperative voiding dysfunction and other complications following a midurethral sling. Am J Obstet Gynecol. 2016 Nov;215(5):656.e1-656.e6. doi: 10.1016/j.ajog.2016.06.010. Epub 2016 Jun 16. PMID 27319367
- [Background] Kleeman S, Goldwasser S, Vassallo B, Karram M. Predicting postoperative voiding efficiency after operation for incontinence and prolapse. Am J Obstet Gynecol. 2002 Jul;187(1):49-52. doi: 10.1067/mob.2002.124841. PMID 12114887
- [Background] Foster RT Sr, Borawski KM, South MM, Weidner AC, Webster GD, Amundsen CL. A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing after transvaginal surgery. Am J Obstet Gynecol. 2007 Dec;197(6):627.e1-4. doi: 10.1016/j.ajog.2007.08.017. PMID 18060956
- [Background] Saint S. Clinical and economic consequences of nosocomial catheter-related bacteriuria. Am J Infect Control. 2000 Feb;28(1):68-75. doi: 10.1016/s0196-6553(00)90015-4. PMID 10679141
- [Background] Dieter AA, Amundsen CL, Visco AG, Siddiqui NY. Treatment for urinary tract infection after midurethral sling: a retrospective study comparing patients who receive short-term postoperative catheterization and patients who pass a void trial on the day of surgery. Female Pelvic Med Reconstr Surg. 2012 May-Jun;18(3):175-8. doi: 10.1097/SPV.0b013e3182544e03. PMID 22543772
- [Background] Pulvino JQ, Duecy EE, Buchsbaum GM, Flynn MK. Comparison of 2 techniques to predict voiding efficiency after inpatient urogynecologic surgery. J Urol. 2010 Oct;184(4):1408-12. doi: 10.1016/j.juro.2010.05.096. Epub 2010 Aug 19. PMID 20727543
- [Background] Ingber MS, Vasavada SP, Moore CK, Rackley RR, Firoozi F, Goldman HB. Force of stream after sling therapy: safety and efficacy of rapid discharge care pathway based on subjective patient report. J Urol. 2011 Mar;185(3):993-7. doi: 10.1016/j.juro.2010.10.050. Epub 2011 Jan 19. PMID 21247598
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Myers EM, Matthews CA, Crane AK, Connolly A, Wu JM, Geller EJ. Two techniques for assessing postoperative voiding function, a randomized trial. Int Urogynecol J. 2017 Oct;28(10):1567-1572. doi: 10.1007/s00192-017-3310-y. Epub 2017 Mar 11. PMID 28285395
- [Background] Goode PS, Locher JL, Bryant RL, Roth DL, Burgio KL. Measurement of postvoid residual urine with portable transabdominal bladder ultrasound scanner and urethral catheterization. Int Urogynecol J Pelvic Floor Dysfunct. 2000;11(5):296-300. doi: 10.1007/s001920070020. PMID 11052565
- [Background] Hakvoort RA, Thijs SD, Bouwmeester FW, Broekman AM, Ruhe IM, Vernooij MM, Burger MP, Emanuel MH, Roovers JP. Comparing clean intermittent catheterisation and transurethral indwelling catheterisation for incomplete voiding after vaginal prolapse surgery: a multicentre randomised trial. BJOG. 2011 Aug;118(9):1055-60. doi: 10.1111/j.1471-0528.2011.02935.x. Epub 2011 Apr 11. PMID 21481147
- [Background] Niel-Weise BS, van den Broek PJ. Urinary catheter policies for short-term bladder drainage in adults. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD004203. doi: 10.1002/14651858.CD004203.pub2. PMID 16034924
- [Background] Kamilya G, Seal SL, Mukherji J, Bhattacharyya SK, Hazra A. A randomized controlled trial comparing short versus long-term catheterization after uncomplicated vaginal prolapse surgery. J Obstet Gynaecol Res. 2010 Feb;36(1):154-8. doi: 10.1111/j.1447-0756.2009.01096.x. PMID 20178542
- [Background] Glavind K, Morup L, Madsen H, Glavind J. A prospective, randomised, controlled trial comparing 3 hour and 24 hour postoperative removal of bladder catheter and vaginal pack following vaginal prolapse surgery. Acta Obstet Gynecol Scand. 2007;86(9):1122-5. doi: 10.1080/00016340701505317. PMID 17712655
- [Background] Kessler TM, Ryu G, Burkhard FC. Clean intermittent self-catheterization: a burden for the patient? Neurourol Urodyn. 2009;28(1):18-21. doi: 10.1002/nau.20610. PMID 18726939
- [Background] Hakvoort RA, Nieuwkerk PT, Burger MP, Emanuel MH, Roovers JP. Patient preferences for clean intermittent catheterisation and transurethral indwelling catheterisation for treatment of abnormal post-void residual bladder volume after vaginal prolapse surgery. BJOG. 2011 Oct;118(11):1324-8. doi: 10.1111/j.1471-0528.2011.03056.x. Epub 2011 Jul 29. PMID 21797960
- [Background] Bickhaus JA, Drobnis EZ, Critchlow WA, Occhino JA, Foster RT Sr. The Feasibility of Clean Intermittent Self-Catheterization Teaching in an Outpatient Setting. Female Pelvic Med Reconstr Surg. 2015 Jul-Aug;21(4):220-4. doi: 10.1097/SPV.0000000000000155. PMID 25679356
- [Background] Parsons BA, Narshi A, Drake MJ. Success rates for learning intermittent self-catheterisation according to age and gender. Int Urol Nephrol. 2012 Aug;44(4):1127-31. doi: 10.1007/s11255-012-0136-x. Epub 2012 Feb 18. PMID 22350836
- [Background] Kowalik U, Plante MK. Urinary Retention in Surgical Patients. Surg Clin North Am. 2016 Jun;96(3):453-67. doi: 10.1016/j.suc.2016.02.004. PMID 27261788
- [Background] Homma Y, Yoshida M, Seki N, Yokoyama O, Kakizaki H, Gotoh M, Yamanishi T, Yamaguchi O, Takeda M, Nishizawa O. Symptom assessment tool for overactive bladder syndrome--overactive bladder symptom score. Urology. 2006 Aug;68(2):318-23. doi: 10.1016/j.urology.2006.02.042. PMID 16904444